CLINICAL TRIAL: NCT04492683
Title: A Phase 2 Study to Evaluate the Sensitivity, Specificity and Safety of DBV1605, a Ready-to-Use Atopy Patch Test for the Diagnosis of Non-Immunoglobulin E Mediated Cow's Milk Allergy in Children
Brief Title: Diagnostic Accuracy and Safety of DBV1605 for the Diagnosis of Non-IgE Mediated Cow's Milk Allergy in Children
Acronym: APTITUDE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: V1605-201
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-12

CONDITIONS: Cow's Milk Allergy
Keywords: Non-IgE mediated CMA
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Disease group (Experimental): One active patch and one control patch applied to subjects with clinical symptoms suggestive of non-IgE mediated CMA
  Interventions: Combination Product: DBV1605
- Control group (Experimental): One active patch and one control patch applied to subjects without any history of allergic disease
  Interventions: Combination Product: DBV1605

INTERVENTIONS:
Combination Product: DBV1605 — Ready-to-use atopy patch test for diagnostic use containing 2 distinct patches:
  * One active patch containing a dry deposit of 180 μg of cow's milk proteins
  * One control patch with the same design as the active patch but devoid of any formulation.

SUMMARY:
Study to assess the diagnostic accuracy (sensitivity, specificity, positive and negative predictive value) of DBV1605 for the diagnosis of non-Immunoglobulin E (IgE) mediated cow's milk allergy (CMA) in children with symptoms suggestive of non-IgE mediated CMA.

ELIGIBILITY:
DISEASE GROUP

Inclusion Criteria:

* Male or female subjects aged > 28 days to ≤ 24 months at Screening Visit
* Subjects with clinical symptoms suggestive of non-IgE mediated Cow's Milk Allergy
* Subjects with any type of diet containing daily products with cow's milk protein (e.g. cow's milk consumption, cow's milk partial elimination, partially hydrolyzed milk) prior to Screening Visit or who have started a cow's milk elimination diet not more than 4 weeks prior to Screening Visit,
* Subjects/parents/guardians who agree to follow a strict cow's milk-free diet and other mammalian milks (such as sheep and goat's milk) as per study requirements.

Exclusion Criteria:

* Subjects with an established diagnosis of non-IgE mediated CMA
* Breast-fed subject at Screening Visit
* Subjects with a convincing history of IgE-mediated CMA
* Subjects on a cow's milk protein-free diet including an AA-based formula or an extensively hydrolyzed formula initiated more than 4 weeks prior to Screening Visit.
* Generalized dermatologic disease (e.g. severe atopic dermatitis, ) extending widely on the skin.
* Any contraindication to a cow's milk challenge

CONTROL GROUP

Inclusion Criteria:

* Male or female subjects aged > 28 days to ≤ 24 months at Screening visit
* Subjects having no medical history of any type of allergy
* Subjects who tolerate at least 200 mL of cow's milk or equivalent dairy foods daily within 4 weeks prior to Screening visit

Exclusion Criteria:

* Subjects with history of persistent gastro-intestinal symptoms
* Exclusively breast-fed subjects at Screening visit

Ages: 29 Days to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of DBV1605 | 48 hours
  Sensitivity and specificity of DBV1605 based on skin reactivity readings after 48 hours will be compared to the results of the DBPCFC in subjects of the disease group.
Diagnostic performance of DBV1605 | 72 hours
  Sensitivity and specificity of DBV1605 based on skin reactivity readings after 72 hours will be compared to the results of the DBPCFC in subjects of the disease group.

SECONDARY OUTCOMES:
Adverse Events (AEs), Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) | Up to day 49

CONTACTS AND LOCATIONS:
Locations (33):
- United States (20):
  - Titan Clinical Research, Phoenix, Arizona
  - University of Arizona Health Science, Tucson, Arizona
  - University of California, Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Eastern Research Inc., Hialeah, Florida
  - Biomedical Research, LLC, Miami, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Allergy Center at Brookstone - Research Department, Columbus, Georgia
  - MedPharmics, LLC - Lafayette, Lafayette, Louisiana
  - Massachusets General Hospital, Boston, Massachusetts
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center (URMC) - Golisano Children's Hospital (GCH), Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University (CWRU) - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Alliance for Multispecialty Research, LLC - New Roy Office, Roy, Utah
- Canada (3):
  - Halton Pediatric Allergy, Burlington, Ontario
  - Hamilton Allergy, Hamilton, Ontario
  - Gordon Sussman Clinical Research Inc., North York, Ontario
- Italy (8):
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - UOC Pediatria ad Indirizzo Gastroenterologico - Ospedale pediatrico Di Cristina, Palermo
  - IRCCS Fondazione Policlinico San Matteo - Pediatria, Pavia
  - Azienda Ospedaliero Universitaria Pisana - Ospedale Santa Chiara, Pisa
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - Università la Sapienza U.O.C di Gastroenterologia, Epatologia e Endoscopia Digestiva Pediatrica, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma, Verona
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Centre of Pediatrics, Vilnius